CLINICAL TRIAL: NCT00300807
Title: A Phase I, Randomized, Double Blind, Placebo-Controlled, Multi-Center Study of the Safety and Virologic Effects of Ascending Single (and Multiple) Doses of XTL6865 in Patients With Chronic Hepatitis C Virus Infection
Brief Title: Study of XTL6865 in Patients With Chronic Hepatitis C Virus Infection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: XTL Biopharmaceuticals (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: XTL2005-16; XTL6865
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Last update posted 2007-03-07 (Estimated); Status verified 2007-03

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Monoclonal Antibody; failed IFN/RBV treatment
MeSH Terms: conditions — Hepatitis C

INTERVENTIONS:
Drug: XTL 6865

SUMMARY:
1. Evaluate the safety, tolerability, and virologic activity of escalating single (and multiple) doses of XTL6865, a mixture (1:1) of two human monoclonal antibodies (HCV-AbXTL68 and HCV-AbXTL65), in patients with chronic hepatitis C virus infection.
2. Assess the pharmacokinetics of XTL6865 in the presence and absence of viral infection.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, and virologic activity of escalating single and multiple doses of XTL6865, a mixture (1:1) of two human monoclonal antibodies (HCV-AbXTL68 and HCV-AbXTL65), in patients with chronic hepatitis C virus infection.

An additional purpose of this study is to assess the pharmacokinetics of XTL6865 in the presence and absence of viral infection.

This study is a randomized, double blind, placebo-controlled, multi-center design of ascending single doses in patients with chronic hepatitis C virus (HCV) infection. In addition to Placebo, the following XTL6865 doses will be administered: 5 mg, 20 mg, 75 mg, 250 mg, 600 mg, 1200 mg, and 2400 mg. No patient will be enrolled in more than one dose level. At each dose level, 3 patients will receive XTL6865 and 1 patient will receive the Placebo. After the single dose infusion, the patients will be followed for 6 weeks.

If certain criteria are met and the safety review of the 1200 mg dose cohort data determines that XTL6865 was safely administered and tolerated at that dose level, the patients in the 600 mg and 1200 mg dose levels are eligible for the multiple dosing phase. Infusions of 600 mgs will be given to 4 eligible patients, one infusion per day, for 5 days. One patient will receive Placebo and 3 patients will receive XTL6865 600 mg. The patients will be followed for 6 additional weeks.

If certain criteria are not met, the 2400 mg dose cohort will be infused. After the safety review has determined that XTL6865 was safely administered and tolerated, the patients in the 1200 mg and 2400 mg dose levels are eligible for the multiple dosing phase. Infusions of 1200 mgs will be given to 4 eligible patients, one infusion per day, for 5 days. One patients will receive Placebo and 3 patients will receive XTL6865 1200 mg. The patients will be followed for 6 additional weeks.

ELIGIBILITY:
Inclusion Criteria:

1. male or female patients between 18 and 65 years of age;
2. female patients must be either postmenopausal, surgically sterile, or non-pregnant and non-lactating and have a negative serum pregnancy test result prior to enrollment into the study. Female patients of childbearing potential (including peri-menopausal women who have had a menstrual period within 1 year) must be using appropriate birth control during the entire duration of the study. Male patients may be either surgically sterile, abstinent, or utilizing a barrier contraceptive method. Abstinence or contraceptive regimen must be maintained during screening, the treatment period and for 6 weeks following the XTL6865 dose;
3. patient has been persistently HCV RNA-positive and remains HCV RNA-positive at screening (patient must have HCV RNA-concentrations which are at least 2 logs above the assay cut-off of 600 IU/mL) and HCV antibody (anti-HCV) positive;
4. patient is negative for human immunodeficiency virus (HIV), hepatitis delta virus (HDV), and has no evidence of chronic hepatitis B virus (HBV) infection (assessed by Hepatitis B surface antigen or HBV DNA in blood within 3 months of Day 1 of the study) or other clinical signs, symptoms, or laboratory abnormalities (e.g. amino transferases) leading to the a diagnosis of current acute Hepatitis B disease;
5. patient is in reasonably good health, as determined by the Investigator based on medical history, physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory tests, except for findings related to their hepatitis C positive status.
6. subject's private physician has been informed of the subject's planned participation in the study;
7. capable of understanding and complying with the protocol, willing to reside in the study unit during the study period and to cooperate fully with the Investigator and site personnel, and must have signed the informed consent document prior to performance of any study-related procedures;
8. infected with HCV genotype 1
9. failed previous treatment for HCV infection with an approved regimen of IFN/RBV or pegylated IFN/RBV. Treatment failure includes both non-response (defined as a patient who did not experience a > 2 log decrease in HCV RNA after 12 weeks of treatment or who failed to clear virus to below the limits of detection after 24 weeks of treatment) or relapse (defined as re-emergence of detectable concentrations of HCV RNA after response to treatment). Treatment must have been discontinued at least 3 months prior to Day 1 of the study.

Exclusion Criteria:

1. liver transplant patients;
2. patients with diabetes and HbA1c at screening of 7% or more;
3. patients who have previously received HCV-AbXTL68;
4. women who are pregnant, lactating, or have a positive serum pregnancy test at screening or positive urine pregnancy test on Day 1 at check-in;
5. patient has hemoglobin < 11 g/dL for women and 12 g/dL for men, platelet count < 50,000 cells/mm3, bilirubin > 3 mg/dL, serum creatinine > 1.5 x normal, INR >1.5 x normal, ALT > 5 x upper limit of normal, or serum albumin < 3.0 g/dL (at screening);
6. patient has a history or evidence of advanced or decompensated liver disease, ascites, encephalopathy, bleeding esophageal varices, hematuria or proteinuria, alcohol or intravenous drug abuse (within <= 1 years), fulminant liver failure, acute hepatitis from any source, periarteritis nodosa, serum sickness, an acute infectious illness, severe psychiatric disorder (including major depression), organic brain disorder, mental retardation, or other clinical conditions or diseases which in the judgment of the Investigator would interfere with the study or confound the results;
7. patient has present active malignancy (except for superficial cancers)
8. past history of pulmonary embolus, deep vein thrombosis, or current therapy with heparin or warfarin;
9. patient has a history of pulmonary hypertension;
10. patient with hypertension that is not, in the investigator's opinion, adequately controlled by medication (DBP > 90 and SBP > 140). In order to assess PK in the fasted state, patients should be able to delay administration of prescribed anti-hypertensive medicine for several hours without anticipating undue risk of medically significant increases in blood pressure. Patient should be on a stable anti-hypertensive regime for at least 30 days prior to screening with no changes in anti-hypertensive medications.
11. patient is currently receiving antiviral therapy for HCV;
12. patient has received IFN/RBV or pegylated IFN/RBV treatment within 3 months of study entry (Day 1);
13. immunomodulatory therapy (eg, systemic corticosteroids or interferon) within 3 months of study entry (Day 1);
14. any patient who does not meet the conditions for prior and concomitant treatments described in Section 6.6 of this protocol;
15. any patient considering or scheduled to undergo any surgical procedure during the study;
16. has taken any other investigational drug during the 30 days prior to screening visit;
17. has donated or lost more than a unit of blood within 30 days prior to screening visit;
18. has any condition(s) that in the Investigator's opinion would: a) warrant exclusion from the study or b) prevent the patient from completing the study;
19. has limited mental capacity or language skills to the extent simple instructions cannot be followed or information regarding adverse events cannot be provided.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2005-10; Study Completion 2007-04

PRIMARY OUTCOMES:
log change in serum concentrations of HCV RNA
change in serum anti-E2 concentrations

CONTACTS AND LOCATIONS:
Overall Officials: John Andrews, PhD, Study Director — XTL Biopharmaceuticals
Locations (5):
- United States (4):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Mt Sinai School of Medicine, New York, New York
  - University Of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Metropolitan Research, Fairfax, Virginia
- Hadassah University Hospital, Jerusalem, Israel